CLINICAL TRIAL: NCT01888965
Title: A Pilot Study of Dovitinib as Maintenance and Adjuvant Therapy in Patients With Colorectal and Pancreas Cancers
Brief Title: Maintenance Dovitinib for Colorectal and Pancreas Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Adverse Event issues.
Sponsor: Georgetown University (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTK1258AUS16T; Pro063 (Other: Georgetown University)
Record Dates: First submitted 2013-06-26; First posted 2013-06-28 (Estimated); Results first posted 2016-07-19 (Estimated); Last update posted 2016-07-19 (Estimated); Status verified 2015-08

CONDITIONS: Colorectal Cancer; Pancreas Cancer
Keywords: Maintenance therapy; Adjuvant Therapy
MeSH Terms: conditions — Colorectal Neoplasms; Pancreatic Neoplasms | interventions — 4-amino-5-fluoro-3-(5-(4-methylpiperazin-1-yl)-1H-benzimidazol-2-yl)quinolin-2(1H)-one

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Dovitinib (Experimental): Dovitinib 500 mg orally daily for 5 days followed by 2 days off (7 day cycles) for up to 2 years
  Interventions: Drug: Dovitinib

INTERVENTIONS:
Drug: Dovitinib — All patients in the study will receive Dovitinib, 500 mg orally daily for 5 days followed by 2 days off (7 day cycles) for up to 2 years.
  If 500 mg is intolerable, 400 mg will be dosed. If 400 mg is intolerable, 300 mg will be dosed
  Other Names: TKI258

SUMMARY:
This study is for patients with stage 4 colon cancer who have had initial chemotherapy or had surgery to remove metastases and patients with pancreas cancer, which has been surgically removed and are receiving adjuvant chemotherapy or is locally advanced and have already received chemotherapy and radiation.

The purpose of this study is to determine the effects of oral dovitinib in patients with advanced stage colorectal and pancreas. Effects include biomarker changes, progression-free survival and safety. Dovitinib will be taken by mouth for 5 days out of every week for up to 2 years.

DETAILED DESCRIPTION:
This is a single institution, nonrandomized, open-label pilot study of dovitinib as maintenance and adjuvant therapy in patients with colorectal and pancreas cancers.

Patient Populations:

Cohort 1: Stage 4 Colon Cancer s/p metastasectomy (Adjuvant cohort)

Cohort 2: Stage 4 Colon Cancer after initial chemotherapy (Maintenance cohort)

Cohort 3: Pancreas Cancer s/p resection and adjuvant chemo (Adjuvant cohort)

Cohort 4: Locally advanced pancreas cancer s/p chemo and radiation (Maintenance cohort)

Each of the 4 cohorts will be accrued independently. 15 patients will be accrued to each cohort. Treatment will begin following the completion of the standard adjuvant or induction therapy. Patients will continue to take dovitinib until they demonstrate progression of disease using standard RECIST criteria, withdraw consent, or experience unacceptable toxicity.

Blood and urine Biomarker studies will be performed on all patients in all cohorts. Samples will be collected at baseline and every 8 weeks for the first 6 months and then every 3 months thereafter, while patients are on study. Blood and urine will be collected and banked for protein, miRNA and metabolomic analysis. Tumor specimens will be taken from patients in maintenance cohorts before and 2 weeks after initiation of dovitinib. All of these samples will be analyzed to determine if biomarkers of benefit and progression can be determined.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a confirmed diagnosis of:

  1. Stage 4 colon cancer either s/p metastasectomy or post-initial chemotherapy or maintenance "standard of care", either involving 5-fluorouracil/leucovorin (5-FU/LV) alone or continual bevacizumab alone. Patients in maintenance cohort must have had 2 consecutive CT scans showing stable disease and not be experiencing significant prior treatment-related toxicity above Grade 1.
  2. Pancreas cancer, either s/p resection and adjuvant chemotherapy or locally advanced pancreas cancer s/p chemotherapy and radiation. Initial chemotherapy or radiation therapy may have been stopped between 2 weeks and 2 months prior to study start, and patients must have recovered from prior treatment related toxicity to grade 1 or less.
* Prior surgery, including tumor resection or metastasectomy must have been performed at least 4 weeks prior to study enrollment.
* No concomitant anti-cancer treatment is allowed
* Age >/= 18 years
* Performance status of 0-1
* Adequate hepatic, bone marrow, and renal function
* Partial thromboplastin time (PTT) must be </= 1.5 x upper normal limit of institution's normal range and INR (International Normalized Ratio) < 1.5.
* Life expectancy >/= 4 months for maintenance cohorts and >/= 6 months for adjuvant cohorts
* Women of childbearing potential must have a negative serum pregnancy test within 14 days prior to initiation of treatment and must not be lactating.
* Subject is capable of understanding and complying with protocol demands and able to sign and date the informed consent

Exclusion Criteria:

* Women of child-bearing potential, who are biologically able to conceive, not employing two forms of highly effective contraception or who are pregnant.
* Women who are breast-feeding
* Fertile males unwilling to use contraception
* Patients with brain metastases or any history of brain metastases
* Patients who have undergone major surgery (e.g., intra-thoracic, -abdominal, or -pelvic) </= 4 weeks prior to starting study treatment or who have not recovered from such therapy
* Patients with a history of pulmonary embolism, or untreated deep vein thrombosis within the past 6 months
* Impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of dovitinib
* The subject has had another active malignancy within the past 5 years except for cervical cancer in situ, in situ carcinoma of the bladder or non-melanoma carcinoma of the skin.
* Patients who have received the last administration of an anticancer therapy including chemotherapy, immunotherapy, hormonal therapy and monoclonal antibodies </= 2 weeks prior to starting the study drug, or who have not recovered from the side effects of such therapy
* Cirrhosis, chronic active hepatitis or chronic persistent hepatitis
* Patients who are currently receiving prasugrel
* No concurrent use of isoniazid, labetolol, trovafloxacin, tolcapone, and felbamate
* No concurrent use of other investigational drugs or antineoplastic therapies.
* Patients with impaired cardiac function or clinically significant cardiac diseases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2013-10; Primary Completion 2014-08 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John L Marshall, MD, Principal Investigator — Georgetown University
Locations (1):
- Georgetown University- Lombardi Cancer Center, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Dovitinib: Dovitinib 500 mg orally daily for 5 days followed by 2 days off (7 day cycles) for up to 2 years
  Dovitinib: All patients in the study will receive Dovitinib, 500 mg orally daily for 5 days followed by 2 days off (7 day cycles) for up to 2 years.
Period: Overall Study
Arm/Group | Dovitinib
Started | 9
Completed | 0
Not Completed | 9
Not completed — Adverse Event | 5
Not completed — Lack of Efficacy | 4

BASELINE CHARACTERISTICS:
Arm/Group | Dovitinib
Number analyzed (Participants) | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 1
Age, Continuous [Median (Full Range); unit: years] | 50.9 [39 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 2
Region of Enrollment [Number; unit: participants]
  United States | 9

OUTCOME MEASURES:

1. Primary Outcome: Biomarker Discovery
Description: Changes in biomarkers from before treatment compared to during or after treatment: expression of pFGFR, pFRS2, pERK, BFGF, VEGF, FGFR1, FGFR2,VEGFR, Ki-67, Asp175, and CA9 in tumor tissue; FGFR, VEGFs, BFGF, PLGF, sVEGFR1/ 2, FGF23, GCSF, PDGF-AB, SDF-1a and SCF levels in serum
Time Frame: 2 years
Population: Data cannot be summarized in the data table because biomarker analysis did not take place after study closure due to insufficient number of samples to yield significant results related to dovitinib administration. Instead, collected samples are stored in our biobank, as consented by all patients, for future Oncological analyses of importance.
Arm/Group | Dovitinib
Number analyzed (Participants) | 0

2. Secondary Outcome: Progression-free Survival
Description: Time in days from study entry until disease progression or death
  Disease progression was defined according to RECIST as at least a 20% increase in the sum of the longest diameter of the target lesions, taking as reference the smallest sum longest diameter recorded since the treatment started, or the appearance of one or more new lesions
Time Frame: 2 years
Population: Patients had either Stage 4 Colon Cancer, post-metastasectomy; Stage 4 Colon Cancer post-initial chemotherapy; Pancreas Cancer, post-resection and adjuvant chemo; or Locally advanced pancreas cancer post-chemo and radiation.
Measure: Median (Full Range); unit: days
Arm/Group | Dovitinib
Number analyzed (Participants) | 9
days | 46 [13 to 287]

3. Secondary Outcome: Safety
Description: Percent of subjects who experience grade 3/ 4 adverse events
Time Frame: 2 years
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Dovitinib
Number analyzed (Participants) | 9
percentage of participants | 56

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Dovitinib
Serious Adverse Events (participants affected / at risk) | 5/9
Other Adverse Events (participants affected / at risk) | 9/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dovitinib (N=9)
Fatigue (General disorders) | 1 (1) — 2 patients = Adjuvant colon cancer; 1 patient = Maintenance colon cancer; 1 patient = Maintenance pancreas cancer
Gastric obstruction (Gastrointestinal disorders) | 1 (1)
neutropenia (Blood and lymphatic system disorders) | 1 (1)
hypertension (Vascular disorders) | 1 (1)
Laryngospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dovitinib (N=9)
diarrhea (Gastrointestinal disorders) | 4 (5)
nausea/vomiting (Gastrointestinal disorders) | 3 (5)
fatigue (General disorders) | 6 (9)
hand-foot syndrome (Skin and subcutaneous tissue disorders) | 1 (1)
rash (Skin and subcutaneous tissue disorders) | 3 (3)
hypertriglycerodemia (Metabolism and nutrition disorders) | 3 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes